CLINICAL TRIAL: NCT03376269
Title: The Effect of Hyperbaric Oxygen on Patients Suffering From Chronic Pain Syndrome (Fibromyalgia) With a History of Psychological Trauma
Brief Title: HBOT Effect on Chronic Pain Syndrome With a History of Psychological Trauma
Acronym: HBOTCSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Director of Sagol Center for Hyperbaric medicine and Research, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202/14
Record Dates: First submitted 2015-04-06; First posted 2017-12-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Fibromyalgia; Chronic Pain Syndrome
Keywords: more than 1 year
MeSH Terms: conditions — Fibromyalgia | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined HBOT/psychotherapy (Active Comparator): combined concurrent intervention of HBOT and creative art psychotherapy.
  Interventions: Biological: HBOT; Behavioral: Psychotherapy
- psychotherapy (Other): single intervention with creative art psychotherapy
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Biological: HBOT — •HBOT of 2 ATA for 90 minutes O2 100%, for 60 treatments
  Arms: Combined HBOT/psychotherapy
Behavioral: Psychotherapy — creative art psychotherapy which includes self drawing and daily diary alongside professional psychotherapy sessions

SUMMARY:
The aim of the study is to evaluate the effect of hyperbaric oxygen therapy (HBOT) on 2 types of patients' population suffering from chronic pain syndrome (Fibromyalgia): patients with history of psychological trauma and patients with history of traumatic brain injury.

DETAILED DESCRIPTION:
This study is a prospective clinical trial. After signing a written informed consent, all patients will be invited to medical evaluation including pain sensitivity examination and a series of questionnaires. In addition, all patients will have chest X-ray, cognitive evaluation, brain MRI and brain Single-photon emission computed tomography (SPECT)

. A second brain MRI, brain SPECT, pain sensitivity evaluation and questionnaires will be done after 3 months of treatment (60 sessions of HBOT). The HBOT procedure will be performed at the Sagol center for hyperbaric medicine and research of Assaf Harofeh Medical Center, Israel.

The following HBOT protocol will be applied for all patients: 12 weeks, 5 times per week, daily administration of 100% O2 for 90 minutes at a pressure of 2 absolute atmospheres (ATA) including 5 minutes air breaks every 30 minutes.

Patients with history of psychological trauma are also being treated with creative art psychotherapy. These patients will be randomly assigned to one of the two groups: (1) single intervention with creative art psychotherapy (psychotherapy group); (2) combined concurrent intervention of HBOT and creative art psychotherapy. Groups 1 will serve as controls during the first 3 months and then will be crossed to get HBOT. Before the cross to the HBOT they will have 2nd full evaluation (questioners and brain imaging).

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age over 18
* Known fibromyalgia (chronic pain syndrome) for more than 1 year

Exclusion Criteria:

* Any past hyperbaric treatment prior to inclusion
* Patients with chest x-ray pathology incompatible with hyperbaric environment
* Patients with middle ear problems
* Patients, who cannot "pump", equals middle ear pressure, effectively
* Patients who suffer from claustrophobia
* Inability or Refusing to sign the Informed Consent Form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity | Change After 3 months
  Using (AlogMed) dolorimeter, pain sensitivity will be examined in 18 trigger points (scale0-18)
Brain microstructure | Change after 3 months
  MRI dynamic tensor imaging sequence will be performed (DTI). Fractional anisotropy (FA) values will be assessed at base line and at 3 months. The changes at 3 months from baseline will be compared
Brain Metabolism | Change after 3 months
  Brain metabolism will be assessed using SPECT at baseline, 3 monthsThe counts for each different Broadmann area values will be calculated. The changes at 3 months from baseline will be compared.

SECONDARY OUTCOMES:
Fibromyalgia Impact on quality of life | Change after 3 months
  Evaluated by Fibromyalgia Impact Questionnaire (FIQ).(scale 0-100)
Short form health survey (sf-36) | Change after 3 months
  Quality of live will be evaluated by Quality of Life RAND Short form 36 questionnaire (SF36).(scale 0-100) higher score means better outcome.
Stress | Change after 3 months t
  Stress will be evaluated using the Perceived stress scale (PSS) questionnaire.(scale 0-51)
Psychological symptoms | Change after 3 months
  Psychological symptoms will be evaluated using Brief Symptom Inventory(BSI) questionnaire.(scale 0-20)
Sensory symptoms | Change after 3 months
  Sensory symptoms will be evaluated using the Sensory Profile questionnaires .
Somatoform Dissociation Questionnaire (SDQ-20) | Change after 3 months
  Dissociation symptoms will be evaluated using the Somatoform Dissociation Questionnaire (SDQ-20).
Childhood trauma psychological effects | Change after 3 months
  Childhood trauma psychological effects will be evaluated using the Childhood Trauma Questionnaire (CTQ) questionnaires.(scale 0-125)

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Derived] Hadanny A, Bechor Y, Catalogna M, Daphna-Tekoah S, Sigal T, Cohenpour M, Lev-Wiesel R, Efrati S. Hyperbaric Oxygen Therapy Can Induce Neuroplasticity and Significant Clinical Improvement in Patients Suffering From Fibromyalgia With a History of Childhood Sexual Abuse-Randomized Controlled Trial. Front Psychol. 2018 Dec 17;9:2495. doi: 10.3389/fpsyg.2018.02495. eCollection 2018. PMID 30618929